CLINICAL TRIAL: NCT00883298
Title: Phase II Study of Bi-Weekly Temozolomide Plus Bevacizumab for Adult Patients With Recurrent Glioblastoma Multiforme
Brief Title: Bi-weekly Temozolomide Plus Bevacizumab for Adult Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Neurosciences, Tucson (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Badruddoja, MD, Neurologist, NeuroOncologist, Center for Neurosciences, Tucson
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVF4514s
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Recurrent Glioblastoma Multiforme; Recurrent Gliosarcoma
Keywords: temozolomide; bevacizumab; Temodar; Avastin; glioblastoma multiforme; gliosarcoma; glioma; GBM; brain tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Experimental): temozolomide plus bevacizumab administered as open label single arm treatment
  Interventions: Drug: temozolomide and bevacizumab

INTERVENTIONS:
Drug: temozolomide and bevacizumab — oral temozolomide 100 mg/m2 days 1-5 & 15-19 every 28-day cycle plus intravenous bevacizumab 10 mg/kg days 1 & 5 every 28-day cycle
  Other Names: Temodar; Avastin

SUMMARY:
Primary objective - to determine the 6-month progression free survival (PFS) of adult patients with recurrent glioblastoma multiforme/gliosarcoma treated with bi-weekly temozolomide plus (Avastin) bevacizumab.

Secondary objectives - to determine radiographic response including specialized MRI sequences, safety and overall survival of adult patients with with recurrent glioblastoma multiforme/gliosarcoma treated with bi-weekly temozolomide plus bevacizumab (Avastin). Additionally, tumor DNA (MGMT) analysis as it relates to survival will be evaluated.

DETAILED DESCRIPTION:
This is a phase II study of the combination of Avastin and temozolomide for patients with recurrent glioblastoma multiforme. Avastin is administered intravenously at a dose of 10 mg/kg on days 1 and 15 every 28 days and temozolomide is administered at a dose of 100 mg/m2 on days 1-5 and 15-19 every 28 days (one cycle). Patients will have a baseline MRI, an MRI scan after the first cycle and every other cycle after that. If there is no evidence of disease progression or unacceptable toxicity, patients will receive one year of therapy. If there is evidence of added benefit (eg: tumor regression), patients can stay on treatment longer than one year, per investigator discretion.

ELIGIBILITY:
Inclusion Criteria:

Patients must have histologically confirmed diagnosis of a glioblastoma multiforme/gliosarcoma and:

* Must have completed at least 2 cycles of adjuvant chemotherapy
* Age > 18 years
* Karnofsky > 60%
* Hematocrit > 29%, ANC > 1,500 cells/dl, platelets > 125,000 cells/dl
* Serum creatinine < 1.5 mg/dl, BUN < 25 mg/dl, serum SGOT and bilirubin < 1.5 times upper limit of normal
* If on corticosteroids, must be on a stable dose for 1 week prior to entry; if clinically possible, the dose should not be escalated over entry dose level
* Signed informed consent approved by the Institutional Review Board prior to study entry
* If sexually active, will take contraceptive measures for the duration of the treatments

Exclusion Criteria:

* Prior toxicity grade ≥ 3 with TMZ
* Prior treatment with bevacizumab
* Female patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control
* Concurrent severe and/or uncontrolled medical disease that could compromise participation in the study
* Acute or chronic liver disease (i.e., hepatitis, cirrhosis)
* Confirmed diagnosis of HIV infection
* Have received investigational drugs less than 4 weeks prior to entry on this study or who have not recovered from the toxic effects of such therapy
* Have received chemotherapy within 2 weeks prior (6 weeks for nitrosourea) to entry on this study, or who have not recovered from the toxic effects of such therapy
* Have received biologic, immunotherapeutic or cytostatic agents within 1 week prior to entry on this study or who have not recovered from the toxic effects of such therapy
* Less than 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant
* Have received radiation therapy within 2 weeks prior to entry on this study or who have not recovered from the toxic effects of such therapy.
* Surgical resection of brain tumor within 4 weeks prior to entry on this study or who have not recovered from side effects of such therapy
* Have had any surgery other than resection of a brain tumor within 4 weeks prior to entry on this study or who have not recovered from side effects of such therapy
* Unwilling to or unable to comply with the protocol
* Evidence of tumor progression within on immediate post radiation brain imaging
* Have not received at least 2 cycles of adjuvant chemotherapy
* Life expectancy of less than 12 weeks
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study

Bevacizumab-Specific Exclusions:

* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
* History of myocardial infarction or unstable angina within 6 months
* History of stroke or transient ischemic attack within 6 months
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture.
* Proteinuria as demonstrated by a UPC ratio greater than or equal to 1.0 at screening
* Known hypersensitivity to any component of bevacizumab

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
6-month progression-free survival. | 6 months

SECONDARY OUTCOMES:
Radiographic response (Gd-MRI) including specialized MRI sequences (T2/FLAIR). | every eight weeks
Incidence and severity of toxicity. | 6 months
Tumor DNA (MGMT) analysis as it relates to survival. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Badurddoja, MD, Principal Investigator — Center for Neurosciences
Locations (1):
- Center for Neurosciences, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No